CLINICAL TRIAL: NCT03114995
Title: Effect of Tailored Use of Tirofiban in Patients With Non-ST-elevation Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention
Brief Title: Tailored Use of Tirofiban for Non-ST-elevation Acute Coronary Syndrome Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Tae-Jin Youn, Professor, Cardiovascular Center, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1111-140-001
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Results first posted 2018-06-08 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Non-ST Elevation Myocardial Infarction
Keywords: Tirofiban; Resistance to antiplatelet agents
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction | interventions — Tirofiban

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (high platelet reactivity - tirofiban) (Experimental): Patients with high platelet reactivity unit (230 or higher) Tirofiban administered dose: 0.4 μg/kg/min continuous infusion for 30 min and then 0.10 μg/kg/min continuous infusion for 12 h
  Interventions: Drug: Tirofiban
- Control C1 (high platelet reactivity - no tirofiban) (No Intervention): Patients with high platelet reactivity unit (230 or higher) Tirofiban was not administered
- Control C2 (low platelet reactivity - no tirofiban) (No Intervention): Patients with low platelet reactivity unit (less than 230) Tirofiban was not administered

INTERVENTIONS:
Drug: Tirofiban
  Other Names: Agrastat
  Arms: Group A (high platelet reactivity - tirofiban)

SUMMARY:
Investigators aimed to test the beneficial effect of tirofiban, a GPIIb/IIIa antagonist, for Non-ST-Elevation Acute Coronary Syndrome Patients who has high resistance to clopidogrel.

DETAILED DESCRIPTION:
Some patients have a poor response to dual antiplatelet therapy (DAPT), and it can result in a poor prognosis after percutaneous coronary intervention (PCI). Devices like Ultegra Rapid Platelet Function Analyzer (VerifyNow®) enable us to quantify platelet reactivity quickly in the catheter laboratory. This means that the poor responders to DAPT can be identified, and the patients' outcomes can be improved by providing additional antiplatelet agents. Tirofiban, a GP IIb/IIIa inhibitor, is a potent antiplatelet agent which is recommended for Non-ST-Elevation acute coronary syndrome (NSTE-ACS) with high risk at presentation. However, its role is not clear for patients stabilized with standard medical treatment but with a poor responsiveness to DAPT.

In this study, Investigators administered tirofiban on top of DAPT to patients with NSTE-ACS undergoing PCI who have a high platelet reactivity (HPR) identified by VerifyNow.

To the best of our knowledge, there are few studies conducted with tirofiban for tailored antiplatelet therapy. Moreover, this is the first randomized study with NSTE-ACS patients for tailored use of tirofiban under the guidance of platelet reactivity.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with NSTE-ACS who need PCI
* loaded with aspirin and clopidogrel at least 6 h before the procedure

Exclusion Criteria:

* thrombocytopenia (platelet count <100,000/μL)
* history of hemorrhagic stroke
* history of ischemic stroke in the recent 2 year
* history of major surgery 6 months prior

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Jin Youn, PhD, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No
not planned

REFERENCES:
- [Result] Patti G, Nusca A, Mangiacapra F, Gatto L, D'Ambrosio A, Di Sciascio G. Point-of-care measurement of clopidogrel responsiveness predicts clinical outcome in patients undergoing percutaneous coronary intervention results of the ARMYDA-PRO (Antiplatelet therapy for Reduction of MYocardial Damage during Angioplasty-Platelet Reactivity Predicts Outcome) study. J Am Coll Cardiol. 2008 Sep 30;52(14):1128-33. doi: 10.1016/j.jacc.2008.06.038. PMID 18804738
- [Result] Hong MK, Mehran R, Dangas G, Mintz GS, Lansky AJ, Pichard AD, Kent KM, Satler LF, Stone GW, Leon MB. Creatine kinase-MB enzyme elevation following successful saphenous vein graft intervention is associated with late mortality. Circulation. 1999 Dec 14;100(24):2400-5. doi: 10.1161/01.cir.100.24.2400. PMID 10595951
- [Result] Fung AY, Saw J, Starovoytov A, Densem C, Jokhi P, Walsh SJ, Fox RS, Humphries KH, Aymong E, Ricci DR, Webb JG, Hamburger JN, Carere RG, Buller CE. Abbreviated infusion of eptifibatide after successful coronary intervention The BRIEF-PCI (Brief Infusion of Eptifibatide Following Percutaneous Coronary Intervention) randomized trial. J Am Coll Cardiol. 2009 Mar 10;53(10):837-45. doi: 10.1016/j.jacc.2008.09.060. PMID 19264239
- [Result] De Labriolle A, Lemesle G, Bonello L, Syed AI, Collins SD, Ben-Dor I, Pinto Slottow TL, Xue Z, Torguson R, Suddath WO, Satler LF, Kent KM, Pichard AD, Lindsay J, Waksman R. Prognostic significance of small troponin I rise after a successful elective percutaneous coronary intervention of a native artery. Am J Cardiol. 2009 Mar 1;103(5):639-45. doi: 10.1016/j.amjcard.2008.10.044. Epub 2009 Jan 17. PMID 19231326
- [Result] Jeremias A, Kleiman NS, Nassif D, Hsieh WH, Pencina M, Maresh K, Parikh M, Cutlip DE, Waksman R, Goldberg S, Berger PB, Cohen DJ; Evaluation of Drug Eluting Stents and Ischemic Events (EVENT) Registry Investigators. Prevalence and prognostic significance of preprocedural cardiac troponin elevation among patients with stable coronary artery disease undergoing percutaneous coronary intervention: results from the evaluation of drug eluting stents and ischemic events registry. Circulation. 2008 Aug 5;118(6):632-8. doi: 10.1161/CIRCULATIONAHA.107.752428. Epub 2008 Jul 21. PMID 18645057
- [Result] Cuisset T, Hamilos M, Sarma J, Sarno G, Wyffels E, Vanderheyden M, Barbato E, Bartunek J, De Bruyne B, Wijns W. Relation of low response to clopidogrel assessed with point-of-care assay to periprocedural myonecrosis in patients undergoing elective coronary stenting for stable angina pectoris. Am J Cardiol. 2008 Jun 15;101(12):1700-3. doi: 10.1016/j.amjcard.2008.02.054. Epub 2008 Apr 18. PMID 18549843
- [Result] Suh JW, Lee SP, Park KW, Lee HY, Kang HJ, Koo BK, Cho YS, Youn TJ, Chae IH, Choi DJ, Rha SW, Bae JH, Kwon TG, Bae JW, Cho MC, Kim HS. Multicenter randomized trial evaluating the efficacy of cilostazol on ischemic vascular complications after drug-eluting stent implantation for coronary heart disease: results of the CILON-T (influence of CILostazol-based triple antiplatelet therapy ON ischemic complication after drug-eluting stenT implantation) trial. J Am Coll Cardiol. 2011 Jan 18;57(3):280-9. doi: 10.1016/j.jacc.2010.08.631. PMID 21232664
- [Derived] Lee W, Suh JW, Park JJ, Yoon CH, Cho YS, Youn TJ, Chae IH. Effect of tailored use of tirofiban in patients with Non-ST-elevation acute coronary syndrome undergoing percutaneous coronary intervention: a randomized controlled trial. BMC Cardiovasc Disord. 2018 Oct 22;18(1):201. doi: 10.1186/s12872-018-0938-6. PMID 30348101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutively enrolled patients who are already stabilized with standard medical treatment and diagnosed with Non-ST elevation acute coronary syndrome (NSTE-ACS) at Seoul National University Bundang Hospital from February 2012 to October 2015
Groups:
- Group A (High Platelet Reactivity - Tirofiban): Patients with high platelet reactivity (HPR) unit (230 or higher) Tirofiban administered dose: 0.4 μg/kg/min continuous infusion for 30 min and then 0.10 μg/kg/min continuous infusion for 12 h
  Tirofiban
- Control C2(Low Platelet Reactivity - no Tirofiban): Patients with low platelet reactivity unit (less than 230) Tirofiban was not administered
Period: Overall Study
Arm/Group | Group A (High Platelet Reactivity - Tirofiban) | Control C1 (High Platelet Reactivity - no Tirofiban) | Control C2(Low Platelet Reactivity - no Tirofiban)
Started | 31 | 31 | 78
Completed | 30 | 30 | 78
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A (High Platelet Reactivity - Tirofiban): Patients with high platelet reactivity unit (230 or higher) Tirofiban administered dose: 0.4 μg/kg/min continuous infusion for 30 min and then 0.10 μg/kg/min continuous infusion for 12 h
  Tirofiban
- Total: Total of all reporting groups
Arm/Group | Group A (High Platelet Reactivity - Tirofiban) | Control C1 (High Platelet Reactivity - no Tirofiban) | Control C2 (Low Platelet Reactivity - no Tirofiban) | Total
Number analyzed (Participants) | 30 | 30 | 78 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (12.8) | 64.5 (12.0) | 62.9 (10.1) | 64.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 11 | 29
  Male | 17 | 25 | 67 | 109

OUTCOME MEASURES:

1. Primary Outcome: Area Under Curve of Serial Cardiac Biomarkers
Description: An area under the curve of serial levels of Troponin I and creatine kinase-MB isoenzyme during 36 hours
Time Frame: 0,6,12,18,24,30,36 hours
Measure: Median (Inter-Quartile Range); unit: Hours*ng/ml
Arm/Group | Group A (High Platelet Reactivity - Tirofiban) | Control C1 (High Platelet Reactivity - no Tirofiban) | Control C2 (Low Platelet Reactivity - no Tirofiban)
Number analyzed (Participants) | 30 | 30 | 78
Hours*ng/ml
  Troponin I | 197.2 [41.5 to 395.7] | 38.0 [8.9 to 313.9] | 121.4 [43.7 to 481.8]
  creatine kinase-MB isoenzyme | 252.5 [48.0 to 470.1] | 92.7 [39.1 to 402.1] | 185.6 [79.8 to 425.3]

2. Secondary Outcome: Percentage of Participants With Periprocedural Myonecrosis
Description: Percentage of participants with periprocedural myonecrosis under the criteria described below.
  When the cardiac biomarkers before the procedure were within the 99th percentile upper reference limit (URL), more than a 5-fold elevation in the URL within 12 hours after percutaneous coronary intervention (PCI) was defined as periprocedural myonecrosis. If the cardiac biomarker level was already above the 99th percentile URL before the procedure and the trend was stationary or decreasing, a ≥20% increase compared to the previous level was considered periprocedural myonecrosis. If the trend was still increasing, the levels at the post-6 hour and 12-hour were compared to determine periprocedural myonecrosis.
Time Frame: 0,6,12,18,24,30,36 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (High Platelet Reactivity - Tirofiban) | Control C1 (High Platelet Reactivity - no Tirofiban) | Control C2 (Low Platelet Reactivity - no Tirofiban)
Number analyzed (Participants) | 30 | 30 | 78
Participants
  Troponin I | 16 | 15 | 26
  creatine kinase-MB isoenzyme | 11 | 10 | 25

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Group A (High Platelet Reactivity - Tirofiban) | Control C1 (High Platelet Reactivity - no Tirofiban) | Control C2 (Low Platelet Reactivity - no Tirofiban)
All-Cause Mortality (participants affected / at risk) | 2/30 | 0/30 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/78
Other Adverse Events (participants affected / at risk) | 4/30 | 1/30 | 8/78
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (High Platelet Reactivity - Tirofiban) (N=30) | Control C1 (High Platelet Reactivity - no Tirofiban) (N=30) | Control C2 (Low Platelet Reactivity - no Tirofiban) (N=78)
Minor bleeding (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 8 (8) — Minor bleeding defined by TIMI criteria

LIMITATIONS AND CAVEATS:
The difference in the distribution of PRU values of subjects estimated from previous literatures leading to small numbers of subjects assigned to the study group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No